CLINICAL TRIAL: NCT04805658
Title: Natural History Study of Retinitis Pigmentosa Type 11
Acronym: ReSa
Status: Active, not recruiting | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Josephine Prener Holtan, Senior Consultant, MD PhD, Oslo University Hospital
Other Study IDs: 179417
Record Dates: First submitted 2021-03-16; First posted 2021-03-18 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2024-04

CONDITIONS: Retinitis Pigmentosa 11; Retinitis Pigmentosa
Keywords: Retinitis; RP; PRPF31
MeSH Terms: conditions — Retinitis Pigmentosa 11; Retinitis Pigmentosa; Retinitis | interventions — Physical Examination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Clinical examinations — Clinical examinations

SUMMARY:
Observational study of patients with retinitis pigmentosa type 11

DETAILED DESCRIPTION:
Natural history study with clinical examination every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of retinitis pigmentosa caused by a disease-causing mutation involving the PRPF31 gene
* Or disease-causing mutation involving the PRPF31 gene without the clinical diagnosis of retinitis pigmentosa

Exclusion Criteria:

* Under 18 years
* Other types of retinitis pigmentosa

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients over the age of 18 with the clinical diagnosis of retinitis pigmentosa type 11 or asymptomatic carriers of the disease.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Progression of disease | 24 mounths
  Retinal function measured by functional and structural testing

CONTACTS AND LOCATIONS:
Overall Officials: Josephine P Holtan, MD, PHD, Principal Investigator — Department of Ophthalmology, Oslo University Hospital
Locations (1):
- Department of Ophthalmology, Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No